CLINICAL TRIAL: NCT01317004
Title: A 6-month, Randomized, Active Comparator, Open-label, Multi-Center Study to Evaluate Patient Outcomes, Safety and Tolerability of Fingolimod (FTY720) 0.5 mg/Day in Patients With Relapsing Remitting Multiple Sclerosis Who Are Candidates for MS Therapy Change From Previous Disease Modifying Therapy (EPOC)
Brief Title: Patients With Relapse Remitting Multiple Sclerosis (RRMS): Candidates for MS Therapy Change
Acronym: EPOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DIT02; 2010-024017-31 (EudraCT Number)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; Fingolimod; Disease Modifying Therapy; TSQM-9
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride; Interferon beta-1a; Glatiramer Acetate; Interferon beta-1b

ARMS (2):
- Fingolimod (Experimental): Patients randomized in this arm received Fingolimod 0.5 mg/day oral capsule for 6 months core period.
  Interventions: Drug: Fingolimod
- Multiple Sclerosis Disease Modifying Treatment (MS DMT) (Active Comparator): Patients randomized in this arm received selected Standard MS DMT such as Interferon beta-1b or Interferon beta-1a or Glatiramer acetate for 6 months.
  Interventions: Drug: Standard MS DMT

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg/day oral capsule
  Other Names: GILENYA™
  Arms: Fingolimod
Drug: Standard MS DMT — Interferon beta 1a or interferon beta 1b or Glatiramer Acetate
  Other Names: Avonex®,; Copaxone®,; Rebif®,; Betaferon®,; Extavia®
  Arms: Multiple Sclerosis Disease Modifying Treatment (MS DMT)

SUMMARY:
The purpose of this study is to evaluate the change in patient-reported treatment satisfaction after 6 months of treatment with fingolimod 0.5mg/day vs. DMT standard of care, using the global satisfaction subscale of the Treatment Satisfaction Questionnaire for Medication (TSQM-9).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with relapsing remitting MS (RRMS) as defined by 2005 revised McDonald criteria.
* Patients who explicitly agree to be assigned to a treatment group that may receive fingolimod or DMT after having been informed about their respective benefits and possible adverse events by the investigator.
* An Expanded Disability Status Scale (EDSS) score of 0-5.5 inclusive.
* Must have received continuous treatment with a single approved and indicated MS DMT for a minimum of 6 months prior to the screening visit. Patients must continue with this MS DMT until the randomization visit.
* Naïve to treatment with fingolimod.

Exclusion Criteria:

* A manifestation of MS other than those defined in the inclusion criteria.
* A history of chronic disease of the immune system other than MS or a known immunodeficiency syndrome.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Patients with uncontrolled diabetes mellitus (HbA1c > 7%).
* Diagnosis of macular edema during Screening Phase.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Renato Turrini, MD, Study Director — Novartis Farma S.p.A.
Locations (15):
- Italy (15):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Ponderano, BI
  - Novartis Investigative Site, Caltanissetta, CL
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Como, CO
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Castelfiorentino, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, San Donato Milanese, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Legnago, VR
  - Novartis Investigative Site, Novara

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual enrollment = 61 because 65 participants were randomized to the study, but only 61 participants received at least one dose of study medication. As such, the participant flow captures the 65 participants randomized and the 61 participants who received drug as the safety set.
Period: Overall Study
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Started | 51 | 14
Safety Set | 50 | 11
Completed | 47 | 5
Not Completed | 4 | 9
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT) | Total
Number analyzed (Participants) | 50 | 11 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.96 (8.69) | 35.82 (7.22) | 37.57 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 8 | 40
  Male | 18 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-reported Treatment Satisfaction
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a psychometric measure of a patient's satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The scores were computed by adding items for each domain, i.e. 1 to 3 for effectiveness, 4 - 6 for convenience and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) X 3 items = 18 for the effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. A positive change from baseline indicates improvement.
Time Frame: baseline, 6 months
Population: Participants from the safety set, who had values at both baseline and month 6, were included in the analysis. The safety set included randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 46 | 10
score on a scale | 19.57 (21.00) | 5.83 (16.47)

2. Secondary Outcome: Change From Baseline in Patient-reported Activities of Daily Living (ADL)
Description: The PRIMUS activity measure is a 15-item assessment used to evaluate patient-reported activities of daily living. The PRIMUS activities score was calculated summing the 15 items, after recoding the responses from 1 - 3 to 0 - 2. Therefore, the total score ranged from 0 - 3-, where high scores were indicative of greater function limitation. A negative change from baseline indicates improvement.
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 49 | 11
score on a scale | 0.19 (2.75) | 0.15 (1.72)

3. Secondary Outcome: Change From Baseline in Patient-reported Fatigue
Description: The fatigue Severity Scale (FSS) is a 9-item scale used to assess fatigue. The FSS score was calculated summing the 9 items of the questionnaire and dividing by the number of non-missing items (each item is based on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree)). A negative change from baseline indicates improvement.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 48 | 11
score on a scale | -0.18 (1.46) | -0.32 (1.21)

4. Secondary Outcome: Change From Baseline in Patient-Reported Effectiveness and Convenience
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 46 | 10
score on a scale
  Effectiveness | 13.53 (28.39) | -1.67 (32.40)
  Convenience | 24.64 (18.28) | 12.78 (25.26)

5. Secondary Outcome: Change From Baseline in Patient-reported Depression
Description: The Beck Depression Inventory Fast Screen (BDI-FS) is a brief, multiple choice, self reported inventory designed to evaluate depression in patients with medical illness. The BDI-FS score was calculated summing the 7 items of the questionnaire. Each item ranged from 0 (not present) to 3 (severe). The total score ranges from 0-3 (minimal depression), 4-8 (mild depression), 9-12 (moderate depression) and 13-21 (severe depression). A negative change from baseline indicates improvement.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 48 | 11
score on a scale | -1.15 (3.59) | -0.12 (3.06)

6. Secondary Outcome: Change From Baseline in Patient-reported Health Related Quality of Life (QOL)
Description: The SF-36v2 is a validated health-related quality of life instrument used in numerous disease states, including MS. It is a self-administered survey that measures 8 domains of health including: physical functioning, role limitations due to physical health, pain, general health, energy/fatigue, social functioning, role limitations due to emotional problems and emotional well-being. Additionally, two summary scale scores can be calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). If half or more questions within a domain were answered, then a score was calculated for that domain. Otherwise, the patient score for that domain was set to missing. If the patient was missing any 1 of the 8 scale scores, then the physical and mental component scores were set to missing. An algorithm was used to create a score from 0 to 100 for each domain score and component score. A positive change from baseline indicates improvement.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 45 | 9
score on a scale
  Physical functioning (n=41,9) | 1.71 (23.07) | -1.11 (20.73)
  Role limitations due to physical health (n=42,9) | 7.14 (37.97) | 5.56 (27.32)
  Pain (n=45,9) | 6.56 (24.32) | 14.44 (15.25)
  General health (n=44,8) | 4.52 (19.43) | 6.25 (14.08)
  Energy/fatigue (n=43,9) | 2.33 (18.81) | 6.48 (33.24)
  Social functioning (n=45,9) | 7.78 (24.90) | 6.94 (25.85)
  Role limitations d/t emotional problems (n=45,9) | 7.04 (41.82) | 3.70 (38.89)
  Emotional well-being (n=43,9) | 2.51 (16.88) | 4.89 (28.13)
  PCS (n=40,8) | 4.52 (18.05) | 7.83 (15.86)
  MCS (n=40,8) | 5.88 (18.21) | 7.28 (24.05)

7. Secondary Outcome: Physician-reported Clinical Global Impression of Improvement (CGI-I)
Description: The CGI-I is a rating scale allowing a physician-reported global evaluation of the subject's improvement over time. The Investigator assessed the subject's clinical change relative to the symptoms at baseline on the CGI-I, a seven-point scale, with rating as follows: 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, 7=Very much worse. A lower score and a negative change from baseline indicate improvement.
Time Frame: 6 months
Population: Participants from the safety set, who had values at month 6, were included in the analysis. The safety set included randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Number analyzed (Participants) | 44 | 9
Percentage of participants
  Much improved | 13.64 | 11.11
  Minimally improved | 36.36 | 11.11
  No change | 47.73 | 66.67
  Minimally worse | 2.27 | 11.11

ADVERSE EVENTS:
Arm/Group | Fingolimod | Multiple Sclerosis Disease Modifying Treatment (MS DMT)
Serious Adverse Events (participants affected / at risk) | 4/50 | 1/11
Other Adverse Events (participants affected / at risk) | 13/50 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=50) | Multiple Sclerosis Disease Modifying Treatment (MS DMT) (N=11)
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Drug ineffective (General disorders) | 1 | 0
Human papilloma virus test positive (Investigations) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=50) | Multiple Sclerosis Disease Modifying Treatment (MS DMT) (N=11)
Lymphopenia (Blood and lymphatic system disorders) | 8 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Injection site reaction (General disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1
Transaminases increased (Investigations) | 4 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.